CLINICAL TRIAL: NCT01198587
Title: A Double Blind Randomized Placebo Controlled Trial of Oral Zinc for Children With Acute Diarrhea in a Developed Nation.
Brief Title: Oral Zinc for the Treatment of Acute Diarrhea in US Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michelle Niescierenko, Clinical Fellow Emergency Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-01-0022
Record Dates: First submitted 2010-09-02; First posted 2010-09-10 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Diarrhea; Gastroenteritis
Keywords: Diarrhea; Gastroenteritis; Zinc Supplementation
MeSH Terms: conditions — Diarrhea; Gastroenteritis | interventions — Zinc Sulfate; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Outpatient Zinc Sulfate (Experimental): Zinc Sulfate
  Interventions: Drug: Zinc Sulfate
- Inpatient Zinc Sulfate (Experimental): Zinc Sulfate
  Interventions: Drug: Zinc Sulfate
- Outpatient Placebo (Placebo Comparator): Placebo oral capsule
  Interventions: Drug: Placebo oral capsule
- Inpatient Placebo (Placebo Comparator): Placebo oral capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Zinc Sulfate — For children ages 6month to 1 year, 12.5mg orally daily for 14 days mixed in 60 mL of fluid.
  For children aged 1 year and above 25mg orally daily for 14 days mixed in 60 mL of fluid.
  Other Names: Treatment
  Arms: Inpatient Zinc Sulfate; Outpatient Zinc Sulfate
Drug: Placebo oral capsule — Effervescent oral capsules with similar taste to treatment drug Zinc Sulfate is provided to each patient randomized to the placebo arms of the study
  Other Names: Placebo
  Arms: Inpatient Placebo; Outpatient Placebo

SUMMARY:
Diarrheal diseases are the third leading cause of mortality in the world, with nearly 2 million deaths annually among children under age 5 years. Several clinical trials of oral zinc supplementation performed in developing country populations have confirmed this nutrient's efficacy in reducing the severity and frequency of diarrhea. The World Health Organization (WHO) has recommended global use of zinc supplementation in all children with diarrhea despite little or no data from trials in industrialized/developed settings. In the United States over 4 million children suffer annually from diarrheal illness. Although mortality is not a significant factor in U.S. cases, 75% of all cases present to medical care resulting in over 200,000 hospitalizations annually for diarrhea. This has significant impact on U.S. healthcare costs, with an average of $391 per outpatient treatment and $2,549 per inpatient treatment spent on each episode of acute diarrheal illness. The goal of this study is to evaluate the effectiveness of oral zinc in decreasing the duration of diarrhea in children treated as outpatients and in decreasing the duration of hospitalization in children treated as inpatients in an industrialized country. The results of this study promise to have a substantial impact on the management of a common pediatric health problem, and could conceivably affect direct and indirect healthcare costs to society.

DETAILED DESCRIPTION:
In developing countries, diarrheal diseases are a leading cause of childhood morbidity and mortality. In the United States an estimated 4.67 million children per year suffer from gastroenteritis with a diarrheal component, impacting the delivery and cost of healthcare. Seventy-five percent of these children are brought to physician care across a range of settings from clinics to emergency departments. Children less than five years of age average 1.3 - 2.5 episodes per year, with 1.4% of those children requiring hospitalization annually. This results in an estimated 209,000 hospitalizations yearly for gastroenteritis. The impact of acute gastrointestinal disease can be felt in the developed world, including the United States, as cost attributed to hospitalization and productivity lost. Attempts at treating gastroenteritis have included Oral Rehydration Solution (ORS), introduced 30 years ago by the WHO, which continues to provide a safe and effective way to maintain hydration during acute illness. ORS, however, does not reduce the volume or frequency of stool output in diarrhea. The anti-diarrheal medication loperamide (Imodium®) was commonly used in children until reports of serious adverse reactions caused its use to fall out of favor. There are no other medications or supplements available to specifically treat the diarrheal component of gastroenteritis and studies have shown that adherence to treatment recommendations regarding fluid therapy is poor because care givers want to reduce duration of illness as opposed to supporting children through the natural course of the disease. The desire to relieve diarrheal symptoms often leads care givers to seek antibiotics during a time of rising antibiotic resistance, as well as other treatments with no proven efficacy.

Zinc is an essential trace element for humans. Its physiologic roles are seen throughout the body as a critical cofactor for enzymatic reactions; most notable are its actions in the gastrointestinal (GI) tract. Zinc is an important component of brush border enzymatic activity which promotes gastrointestinal absorption, it regulates water/electrolyte transport at the cellular level, and it enhances the repair of the intestinal mucosa by bolstering immune function. Over the past 10-15 years, there have been more than a dozen randomized controlled trials of zinc supplementation performed in children living in developing countries that have reported improvements in the duration and severity of diarrhea when compared to placebo in a variety of in- and outpatient settings. The majority of zinc trials were conducted in countries at high risk of zinc deficiency, but those conducted at medium risk showed similar effect on duration and severity. When stratified across all nutritional groups based on serum zinc levels a significant effect was seen compared to placebo despite baseline zinc level, with no occurrence of serious adverse reaction in any group. Given these results, the WHO has endorsed zinc supplementation for all children with acute diarrhea, despite the lack of data from similarly designed studies in industrialized/developed settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children with non-bloody diarrhea illness defined as loose or watery stools
* Symptoms must be present for greater than 24 hours but less than 72 hours.
* Comorbid conditions including; Asthma, Gastroesophageal reflux (unless followed by a Gastroenterologist), Mild speech, language, motor delays, Benign heart murmurs, Isolated atrial septal defect (ASD) or ventricular septal defect (VSD), Epilepsy (unless developmentally delayed), Children born Prematurely between 33-37 weeks without long term sequelae, Repaired tetralogy of fallot (no cardiac issues for >6 months), Diabetes may be enrolled in the study.

Exclusion Criteria:

* Children with symptoms less than 24 hours
* Children with symptoms greater than 24 hours
* Failure to thrive
* G or J tube
* Major surgery within last 3 months
* Minor surgery (tonsillectomy, ear tubes, skin lesion removals etc) within last 1 month
* Followed by GI service for any reason (crohns, ulcerative colitis, constipation)
* Developmental delay, patient >1 year behind milestones
* Current brain tumor
* Currently being treated for cancer or in remission < 6 months
* Intussuception
* Antibiotics in the last 14 days or currently taking antibiotics for any reason
* Autism
* Children born premature <33 weeks
* Cystic Fibrosis
* Major congenital Heart Disease (any disease where child's baseline oxygen saturations <93%)
* Short Gut
* Liver disease
* History of bowel resection

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Niescierenko, MD, Principal Investigator — Boston Children's Hospital; Richard Bachur, MD, Principal Investigator — Boston Children's Hospital; Christopher Duggan, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were screened from the emergency department to identify patient meeting study enrollment criteria
Groups:
- Outpatient Zinc Sulfate: Outpatients with diarrhea will be randomized to either zinc or placebo to assess the effect on duration of diarrhea.
  Zinc Sulfate: For children ages 6month to 1 year, 12.5mg orally daily for 14 days mixed in 60 mL of fluid.
  For children aged 1 year and above 25mg orally daily for 14 days mixed in 60 mL of fluid.
- Inpatient Zinc Sulfate: Patients admitted to the hospital with diarrhea and dehydration will be randomized to zinc or placebo, duration of hospitalization will be assessed.
  Zinc Sulfate: For children ages 6month to 1 year, 12.5mg orally daily for 14 days mixed in 60 mL of fluid.
  For children aged 1 year and above 25mg orally daily for 14 days mixed in 60 mL of fluid.
- Outpatient Placebo: Patient discharged randomized to Placebo Oral Capsule
- Inpatient Placebo: Hospitalized patients randomized to Placebo oral capsule
Period: Overall Study
Arm/Group | Outpatient Zinc Sulfate | Inpatient Zinc Sulfate | Outpatient Placebo | Inpatient Placebo
Started | 31 | 5 | 30 | 5
Completed | 23 | 5 | 21 | 5
Not Completed | 8 | 0 | 9 | 0
Not completed — Lost to Follow-up | 8 | 0 | 9 | 0

BASELINE CHARACTERISTICS:
Population: Overall low number of inpatients with diarrhea meeting the study enrollment criteria of being otherwise healthy
Groups:
- Outpatient Zinc Sulfate: Outpatients with diarrhea will be randomized to Zinc Sulfate
  Zinc Sulfate: For children ages 6month to 1 year, 12.5mg orally daily for 14 days mixed in 60 mL of fluid.
  For children aged 1 year and above 25mg orally daily for 14 days mixed in 60 mL of fluid.
- Inpatient Zinc Sulfate: Patients admitted to the hospital with diarrhea and dehydration will be randomized to zinc Sulfate
  Zinc Sulfate: For children ages 6month to 1 year, 12.5mg orally daily for 14 days mixed in 60 mL of fluid.
  For children aged 1 year and above 25mg orally daily for 14 days mixed in 60 mL of fluid.
- Outpatient Placebo: Outpatients with diarrhea will be randomized to Placebo oral capsule
- Inpatient Placebo: Patients admitted to the hospital with diarrhea and dehydration will be randomized to Placebo oral capsule
- Total: Total of all reporting groups
Arm/Group | Outpatient Zinc Sulfate | Inpatient Zinc Sulfate | Outpatient Placebo | Inpatient Placebo | Total
Number analyzed (Participants) | 31 | 5 | 30 | 5 | 71
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 2.3 [1.1 to 3] | 2.9 [2 to 3.1] | 2 [0.98 to 2.6] | 3.6 [1.4 to 5.1] | 2.7 [1.52 to 3.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 12 | 2 | 30
  Male | 18 | 2 | 18 | 3 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 5 | 30 | 5 | 71

OUTCOME MEASURES:

1. Primary Outcome: Duration of Diarrhea in Acute Diarrheal Illnesses in a Developed Nation While Taking Zinc or Placebo.
Description: Patients symptoms will be assessed to identify the duration of diarrhea between zinc and placebo groups before it becomes chronic diarrhea which by definition lasts longer than 14 days. Outcome of all patients in study will be assessed at study conclusion.
Time Frame: 14 days
Population: The study failed to enroll sufficient inpatients due to the low hospitalization rate in the US for children who are otherwise healthy with diarrhea All patients were analyzed separately by arm and then again together for overall severity of diarrhea
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Inpatient Zinc Sulfate: Patients admitted to the hospital with diarrhea and dehydration will be randomized to zinc sulfate.
  Zinc Sulfate: For children ages 6month to 1 year, 12.5mg orally daily for 14 days mixed in 60 mL of fluid.
  For children aged 1 year and above 25mg orally daily for 14 days mixed in 60 mL of fluid.
- Inpatient Placebo: Hospitalized patients with diarrhea and dehydration will be randomized to placebo oral capsule
Arm/Group | Outpatient Zinc Sulfate | Inpatient Zinc Sulfate | Outpatient Placebo | Inpatient Placebo
Number analyzed (Participants) | 23 | 5 | 21 | 5
Hours | 73 (77.8) | 72 (78.7) | 48 (52.6) | 76.8 (81.2)
Statistical Analysis 1: Comparison: Inpatient Zinc Sulfate vs Inpatient Placebo; Test type: Superiority; p = 0.88, Log Rank
Statistical Analysis 2: Comparison: Outpatient Zinc Sulfate vs Outpatient Placebo; Test type: Superiority; p = 0.19, Log Rank

2. Secondary Outcome: Examine the Potential Cost Benefits of Supplementation With Zinc in Reducing Number of Daycare Days Not Attended and Work Days Lost by Parents
Time Frame: over the 14 day symptom monitoring period
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Outpatient Placebo: Outpatients with diarrhea randomized to placebo oral capsules
- Inpatient Placebo: patients with diarrhea and dehydration hospitalized and randomized to placebo oral capsule
Arm/Group | Outpatient Zinc Sulfate | Inpatient Zinc Sulfate | Outpatient Placebo | Inpatient Placebo
Number analyzed (Participants) | 23 | 5 | 21 | 5
Hours
  Daycare Days Lost | 95.3 (9.3) | 29.5 (27.5) | 93.7 (9.6) | 29.5 (27.5)
  Work Days Lost | 93.5 (9.3) | 34 (27.5) | 93.5 (9.6) | 21 (26)

3. Secondary Outcome: Assess Parent Reporting Reliability Comparing Survey Responses to Phone Interview.
Description: Kappa inter-rater reliability measurement was done to analyze the agreement between the phone call data with parents reporting the number of episodes of diarrhea per day were compared to the written symptom charts where parents recorded the number of episodes of diarrhea per day. The inter-rater reliability ranges from 0 to 1 with scores of 0-0.2 = poor agreement, 0.2-0.4 = fair agreement, 0.4-0.6 = moderate agreement, 0.6-0.8 = good agreement and 0.8-1 = very good agreement
Time Frame: agreement over the 14 day follow up period
Population: All patients enrolled in the study
Measure: Number; unit: kappa statistic
Groups:
- Outpatient Placebo: Outpatients with diarrhea randomized to placebo oral capsule
Arm/Group | Outpatient Zinc Sulfate | Inpatient Zinc Sulfate | Outpatient Placebo | Inpatient Placebo
Number analyzed (Participants) | 23 | 5 | 21 | 5
kappa statistic | 0.84 | 0.84 | 0.84 | 0.84

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected for each patient for their 28 day study period. The trial was conducted from November 1 2010 to May 25 2014. The primary completion date of the trial was May 15th 2014 and the study completion date was May 25th 2014.
Arm/Group | Outpatient Zinc Sulfate | Inpatient Zinc Sulfate | Outpatient Placebo | Inpatient Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/5 | 0/21 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/5 | 0/21 | 0/5
Other Adverse Events (participants affected / at risk) | 2/23 | 0/5 | 2/21 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Zinc Sulfate (N=23) | Inpatient Zinc Sulfate (N=5) | Outpatient Placebo (N=21) | Inpatient Placebo (N=5)
Surgical abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 — Disorder requiring abdominal surgery occurred
Hospitalization after starting the study protocol within 14 days (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patients will be assess to identify if the admission is related (for example a motor vehicle accident would be unrelated) and if the reason for admission could be related to the study medication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Zinc Sulfate (N=23) | Inpatient Zinc Sulfate (N=5) | Outpatient Placebo (N=21) | Inpatient Placebo (N=5)
discontinued due to vomiting/tast (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 | 0 — Drug stopped by parent/guardian due to taste or vomiting (difficult to distinguish between the two in young children)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes